CLINICAL TRIAL: NCT04538079
Title: Non-invasive Objective Assessment of Hemodynamics in Preterm Neonates - the NOAH Study
Brief Title: Non-invasive Objective Assessment of Hemodynamics in Preterm Neonates
Acronym: NOAH
Status: Terminated | Type: Observational
Why Stopped: End of funding period
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Professor, University College Cork
Other Study IDs: ED001/19UCC
Record Dates: First submitted 2020-03-05; First posted 2020-09-03 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Hypotension and Shock; Hypoperfusion; Hemodynamic Instability; Intraventricular Hemorrhage; Cardiac Function; Circulatory Transition
Keywords: objective hemodynamic multimodal Monitoring; premature preterm infant
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Feasibility/Accuracy/Reproducibility: The first 20 participants will be analysed for feasibility and the first 40 ECHOs for accuracy/reproducibility of non-invasive Cardiac Output Monitoring with ECHO as reference Method.
  Interventions: Device: Multimodal objective non-invasive Monitoring
- Prediction of Circulatory Failure: Together with the Feasibility/Accuracy/Reproducibility Cohort this group's results will be analysed for prediction of circulatory failure defined as an ultrasound abnormality (IVH grade 3 - 4) or death within the first two weeks of life.
  Interventions: Device: Multimodal objective non-invasive Monitoring

INTERVENTIONS:
Device: Multimodal objective non-invasive Monitoring — Multimodal objective non-invasive monitoring including cerebral oxygenation (NIRS), pulse oximetry with Pulsatility Index (PI) and non-invasive Cardiac Output Monitoring will be recorded but not used for clinical decision making. 2 ECHOs will be performed (one within the first 24h, one in the 2nd 24 hours after birth)

SUMMARY:
Study type: Prospective Observational trial Study design: Longitudinal Population: Preterm newborns <32 weeks gestational age Hypothesis: The inclusion of non-invasive physiological measures of cardiac output, peripheral perfusion and brain oxygenation (NIRS) for preterm neonates is feasible and reveals additional information on the hemodynamic status compared to blood pressure alone. These measurements can improve the ability to rapidly identify those infants who might benefit from intervention and are correlated with short term clinical outcomes.

DETAILED DESCRIPTION:
Understanding neonatal hemodynamics is key to neonatal care. Despite decades of research, uncertainty continues as to how best assess impaired hemodynamics.

Hypotension defined by a low Mean Arterial Blood Pressure (MABP) remains a common issue in preterm infants, affecting up to 30% of extremely preterm infants.

It is common to focus only on MABP thus neglecting the complex and dynamic (patho)physiology that may be present in newborn infants. Providing sufficient cellular oxygenation is the primary task of the circulatory system and different factors may compromise it. In this prospective observational study the investigators will examine various forms of objective non-invasive continuous hemodynamic monitoring methods in very preterm infants

1. For feasibility of non-invasive CO measurement (first 20 patients)
2. For reproducibility and correlation of this measurement and ECHOcardiography (first 40 echocardiographic examinations)
3. For prediction of therapy response.
4. For correlation with clinical definitions of hypotension/hypoperfusion
5. For prediction of later clinical problems/complications of prematurity and impaired hemodynamic status.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of 23 weeks 0 days to 31 weeks 6 days
* NIRS/non-invasive Cardiac Output - device available
* Parental Informed Consent

Exclusion Criteria:

* Congenital anomalies
* Major cardiac defects
* Hydrops
* Parents decline to consent to the study

Ages: 1 Minute to 20 Hours | Sex: All
Age Groups: Child
Study Population: Preterm Neonates born at a gestational age of 23 weeks 0 days to 31 weeks 6 days.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-11-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Adverse Outcome of Circulatory Failure | 14 days
  Correlation of clinical, laboratory, conventional and multimodal non-invasive monitoring and/or a combination of variables with ultrasound abnormality (IVH grade 3 - 4/any IVH) or death within the first two weeks of life.

SECONDARY OUTCOMES:
Feasibility of non-invasive Cardiac Output Monitoring and Pulsatility Index | 48 hours
  The proportion of infants in whom a continuous recording of non-invasive cardiac output (CO) and perfusion index (PI) analysis was obtained for at least 24 hours during the first 48 hours after birth with a good signal quality index
Reproducibility of absolute left ventricular cardiac output estimated by echocardiography compared to cardiac output estimated by non-invasive Cardiac Output Monitoring | 48 hours
  Reproducibility of cardiac output estimates by non-invasive Cardiac Output compared to echocardiographic examinations will be performed using absolute left ventricular output [mL/min]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Reproducibility of left ventricular cardiac output indexed to bodyweight estimated by echocardiography compared to cardiac output estimated by non-invasive Cardiac Output Monitoring | 48 hours
  Reproducibility of cardiac output estimates by non-invasive Cardiac Output compared to echocardiographic examinations will be performed using left ventricular output indexed to bodyweight [mL/kg bodyweight/min]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Reproducibility of left ventricular stroke volume estimated by echocardiography compared to cardiac output estimated by non-invasive Cardiac Output Monitoring | 48 hours
  Reproducibility of left ventricular stroke volume estimates by non-invasive Cardiac Output compared to echocardiographic examinations will be performed using stroke volume [mL]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Reproducibility of absolute right ventricular cardiac output indexed to bodyweight estimated by echocardiography compared to cardiac output estimated by non-invasive Cardiac Output Monitoring | 48 hours
  Reproducibility of absolute cardiac output estimated by non-invasive Cardiac Output Monitoring compared to echocardiographic examinations will be performed using right ventricular output [mL/min]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Reproducibility of right ventricular cardiac output indexed to bodyweight estimated by echocardiography compared to estimation by non-invasive Cardiac Output Monitoring | 48 hours
  Reproducibility of relative right ventricular cardiac output estimates by non-invasive Cardiac Output Monitoring compared to echocardiographic examinations will be performed using right ventricular output indexed to bodyweight [mL/kg bodyweight/min]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Reproducibility of left ventricular systolic time interval ratio estimated by non-invasive Cardiac Output Monitoring compared to echocardiography | 48 hours
  Reproducibility of left ventricular systolic time interval ratio estimates by non-invasive Cardiac Output-Monitoring and echocardiographic examinations will be compared using left ventricular pre-ejection period to left ventricular output time ratio [no unit]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Reproducibility of absolute superior vena cava flow estimated by non-invasive Cardiac Output Monitoring compared to estimation by echocardiography | 48 hours
  Cardiac output estimates of non-invasive Cardiac Output-Monitoring and echocardiographic examinations will be compared using absolute superior vena cava flow [mL/min]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Reproducibility of superior vena cava flow indexed to bodyweight estimated by non-invasive Cardiac Output Monitoring compared to estimation by echocardiography | 48 hours
  Cardiac output estimates of non-invasive Cardiac Output-Monitoring and echocardiographic examinations will be compared using superior vena cava flow indexed to bodyweight [mL/kg bodyweight/min]. The Investigators will use Bland-Altman analysis (Bland-Altman plots, Repeatability coefficient. Repeatability Index will be used for between parameter comparison.
Correlation of non-invasive Cardiac Output Monitoring with echocardiography | 48 hours
  CO-Monitoring and echocardiography will be analysed for correlation using correlation coefficient analysis pairwise for left and right ventricular output indexed to bodyweight [mL/kg bodyweight/min], left ventricular pre-ejection period to left ventricular output time ratio and Superior Vena Cava-flow indexed to bodyweight [mL/kg bodyweight/min].
Prediction of response to volume/red-blood cell transfusion by Corrected Flow Time estimated with non-invasive Cardiac Output Monitoring | 48 hours
  Treatment Responsiveness (Volume and/or red blood cells responsiveness) using trend analysis within Corrected Flow Time (FTC [ms]) for volume responsiveness including a receiver operating characteristic analysis for infants who received volume and/or red blood cells during the study period. (Comparison of 20min mean as baseline before, during and 20min after treatment. Response is defined as normalization of the above mentioned physiological parameters within 20 minutes after receiving treatment.
Prediction of response to volume/red-blood cell transfusion by St roke Volume Variation estimated with non-invasive Cardiac Output Monitoring | 48 hours
  Treatment Responsiveness (Volume and/or red blood cells responsiveness) using trend analysis within Stroke Volume Variation (SVV) for volume responsiveness including a receiver operating characteristic analysis for infants who received volume and/or red blood cells during the study period. (Comparison of 20min mean as baseline before, during and 20min after treatment. Response is defined as normalization of the above mentioned physiological parameters within 20 minutes after receiving treatment.
Prediction of Prediction of response to inotropes by non-invasive Cardiac Output Monitoring response to therapy by non-invasive Cardiac Output Monitoring | 48 hours
  Treatment Responsiveness (Inotrope) using trend analysis within left ventricular cardiac output indexed to bodyweight [ml/kg bodyweight/min] for inotrope responsiveness including a receiver operating characteristic analysis for infants who received inotropes during the study period. (Comparison of 20min mean as baseline before, during and 20min after initiation of inotrope treatment. Response is defined as normalization of the above mentioned physiological parameters within 20 minutes after receiving treatment.
Correlation with definitions of hypotension | 48 hours
  Correlation of multimodal non-invasive monitoring with commonly used definitions of hypotension (Mean Arterial Blood Pressure MABP below 30mmHG and/or MABP below gestational age in weeks)

OTHER OUTCOMES:
Burden of clinical suspicion indicating Circulatory Insufficiency | 48 hours
  Onset and duration of clinical suspicion of Circulatory Insufficiency in clinical examination (i.e. skin colour, increased capillary refill time>3seconds) as documented in the clinical charts.
Burden of Laboratory parameters indicating Circulatory Insufficiency | 48 hours
  Onset and duration of circulatory insufficiency indicated by laboratory parameters (metabolic acidosis with pH<7,2 Lactate>3mmol/L not explainable by intrapartum complications)
Burden and Onset of Hypotension indicating Circulatory Insufficiency | 48 hours
  Time spend with Mean Arterial Blood Pressure (MABP) below 30mmHG and/or MABP below gestational age in weeks
Burden of Cerebral Oxygenation indicating Circulatory Insufficiency | 48 hours
  Time spend wit cerebral regional tissue Saturation (rcStO2) below a value of 60% and/or rcStO2/fraction of tissue oxygen extraction (rcFtO2E) below the infants median value-5%
Burden of Low Cardiac Output indicating Circulatory Insufficiency | 48 hours
  Time spend with Cardiac Output in the lower quartile of the Cohort.
Burden of impaired cerebral Autoregulation | 48 hours
  Time spend with pressure passivity of cerebral regional tissue oxygenation (MABP and or Pulse Pressure to rcStO2/rcFtO2E). Adjusted mutual information and transfer entropy will be used to quantify coupling between MABP or pulse pressure and rcStO2 or rcFtO2E.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene M Dempsey, MD, Principal Investigator — UCC
Locations (1):
- Neonatal Unit Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No